CLINICAL TRIAL: NCT01933347
Title: Third-line Treatment of Gefitinib in NSCLC Patients Who Had Received First-line Gefitinib With EGFR 19del/L858R Mutation and Tumor Progression After the Second-line Chemotherapy: a Single-arm, Prospective and Multi-center Study
Brief Title: Third-line Treatment of Gefitinib in NSCLC Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Guangdong Association of Clinical Trials (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CTONG1304
Record Dates: First submitted 2013-08-28; First posted 2013-09-02 (Estimated); Last update posted 2020-02-06 (Actual); Status verified 2018-04

CONDITIONS: Non Small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Gefitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Gefitinib 250mg/d (Experimental): Subjects will receive the oral administration of gefitinib 250mg/d until the tumor progression, perform scheduled visits in investigational sites at interview day and complete related examinations during follow-up period.
  Interventions: Drug: Gefitinib

INTERVENTIONS:
Drug: Gefitinib — Subjects will receive the oral administration of gefitinib 250mg/d until the tumor progression.
  Other Names: Iressa

SUMMARY:
The purpose of this study is to evaluate the disease control rate (DCR) of gefitinib as third-line retreatment in stage IIIB/IV NSCLC with EGFR 19del/L858R positive mutation patients who had benefited from first-line gefitinib treatment with EGFR 19del/L858R positive mutation and tumor progression after the second-line chemotherapy

DETAILED DESCRIPTION:
* Primary Study Objective: To evaluate the disease control rate (DCR) of gefitinib as third-line retreatment in stage IIIB/IV NSCLC with EGFR 19del/L858R positive mutation patients who had benefited from first-line gefitinib treatment with EGFR 19del/L858R positive mutation and tumor progression after the second-line chemotherapy
* Secondary Study Objectives: To evaluate objective response rate (ORR), progressive-free survival (PFS), overall survival(OS) and quality of life (QoL) of gefitinib as third-line retreatment in NSCLC patients To evaluate the safety of gefitinib as third-line treatment in NSCLC patients
* Exploratory analyses: To dynamically monitor EGFR mutation status and explore the relationship with clinical outcome

ELIGIBILITY:
Inclusion Criteria:

1. The subject or legal guardian could understand and sign informed consent form.
2. Male or female aged 18 years or older;
3. Subjects were diagnosed with stage IIIB or IV NSCLC before starting the first dose of gefitinib third-line treatment;
4. EGFR exon 19 deletion or exon 21 L858R substitution mutation confirmed;
5. ECOG performance status 0-2;
6. Life expectancy of at least 12 weeks or longer;
7. Has at least one measureable lesion by RECIST 1.1;
8. NSCLC of enrolled subjects previously progressed after first-line gefitinib treatment (PFS ≥ 6 months) and progressed again after second-line chemotherapy (not limited for chemotherapy regimen, ≥ 4 cycles of chemotherapy). Investigator considers adopting third-line gefitinib retreatment;
9. Criteria for laboratory examinations:

   * Total bilirubin (TB) ≤ 1.5 times upper limit of normal
   * Aspartate aminotransferase(AST), alanine aminotransferase (ALT) ≤2 times upper limit of normal; for subjects with hepatic metastasis, AST,ALT≤ 5 times upper limit of normal
   * Creatinine clearance≥45ml/min

Exclusion Criteria:

1. Known severe hypersensitivity to gefitinib or any ingredients of the product;
2. Patients with prior exposure to agents directed at the EGFR axis except gefitinib (e.g. erlotinib, cetuximab, trastuzumab) ;
3. Pre-existing interstitial lung disease or pulmonary fibrosis evidenced by CT scan at baseline;
4. Neutrophil count <1.0×109/L or platelet count <50×109/L;
5. Severe infection, uncontrolled systemic disease (e.g cardiopulmonary insufficiency, fatal arrhythmias, hepatitis, etc);
6. Pregnancy or breast-feeding;
7. Women of childbearing age refuse to take adequate contraception measures during gefitinib treatment
8. Subjects with other malignant tumors combined;
9. Known or suspected brain metastases or spinal cord compression, unless treated with surgery and/or radiation and stable without steroid treatment for at least 4 weeks prior to the first dose of study medication;
10. Subjects are unable to take medications orally or have digestive malabsorption;
11. Investigators consider subjects should not be involved in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2014-04-07 (Actual); Primary Completion 2017-04-10 (Actual); Study Completion 2018-04-10 (Actual)

PRIMARY OUTCOMES:
Disease Control Rate (DCR) | week 8

SECONDARY OUTCOMES:
objective response rate (ORR), progressive-free survival (PFS), overall survival(OS) | until the death of last subject or 2 years after enrollment

CONTACTS AND LOCATIONS:
Overall Officials: Yong Song, Ph.D, Principal Investigator — Nanjing PLA General Hospital
Locations (1):
- Nanjing General Hospital of Nanjing Military Command, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No